CLINICAL TRIAL: NCT02889575
Title: Prospective Multicenter Study to Assess the Predictive Value of PIIINP and Urinary NGAL in Renal Function Recovery During Acute Tubular Necrosis
Brief Title: Predictive Value of PIIINP and Urinary NGAL in Renal Function Recovery
Acronym: PIIINP-NGAL
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PROG/11/59
Record Dates: First submitted 2016-08-24; First posted 2016-09-05 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-08

CONDITIONS: Acute Renal Failure; Acute Kidney Tubular Necrosis; Chronic Kidney Failure
MeSH Terms: conditions — Acute Kidney Injury; Kidney Tubular Necrosis, Acute; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Acute Renal Failure (ARF) is defined by a severe, and usually reversible, glomerular filtration rate decreasing. Acute Tubular Necrosis (ATN) remain the major cause of ARF involving distress and destruction of tubular cells. This specific typology of ARF may evolve toward Chronic Renal Failure (CRF) concretizing a major public health issue.

Predict the progression of ARF towards CRF appears essential. The investigators believe that the PIIINP and urinary NGAL biomarkers may constitute robust biomarkers of progression risk towards CRF.

DETAILED DESCRIPTION:
Acute Renal Failure (ARF) is defined by a severe, and usually reversible, glomerular filtration rate decreasing. Beside its frequency, ARF may be associated with severe prognostic. Thus, patient admitted in ICU and suffering of ARF requiring dialysis, had a higher risk of mortality up to 50%.

Tubulointerstitial nephropathies, particularly Acute Tubular Necrosis (ATN) remain the major cause of ARF, representing 45-50% of cases. The ATN is due to suffering and destruction of tubular cells which are very sensitive to ischemia-reperfusion lesions because tubular reabsorption functions require significant and constant energy intake. However, ATN represents a relatively homogeneous group in terms of acute kidney disease typology. Homogeneity and significant frequency compels ATN as an optimal model to study function recovery after ARF.

ARF constitutes a major public health issue. Actually, incidence of Chronic Renal Failure (CRF) after an ARF, due to ATN, is estimated between 19% and 31%. In addition 12.5% of patients with specific ARF presentation immediately reach End-stage Renal Disease (ESRD), and the occurrence of ARF requiring dialysis, triples the risk of chronic renal support.

Therefore, predict the progression of ARF towards CRF appears essential.

At this time, the investigators currently lack of reliable biomarkers to predict such progression. This pejorative kidney development is due to the persistence of intrarenal inflammation, rapid development of interstitial fibrosis and deficiency in tubular restoration. It involves complex mechanisms of inflammatory response, and vascular and tubular remodeling.

Two promising biomarkers of renal fibrosis, ARF occurrence and CRF progression risk appear in recent years: the Procollagen III N-terminal peptide (PIIINP) and the neutrophil gelatinase associated lipocalin (NGAL). The investigators believe that the PIIINP and urinary NGAL may constitute robust biomarkers of progression (or not) towards CRF in ARF context. Firstly, PIIINP is a good reflection of fibrosis process inside the kidney. Secondarily, NGAL is a marker of renal tubule remodeling after renal aggression. The combination of these two biomarkers could therefore efficiently reflect the balance tubular fibrosis/restoration and may allow optimal prediction of renal function recovery.

The investigators hypothesize that these two biomarkers may be used to assess the risk of CRF progression during ARF in ATN context.

ELIGIBILITY:
Inclusion Criteria:

* off-age patient.
* ATN diagnosis based on 1) typical clinical environment (sepsis, nephrotoxicity...) 2) 50% decrease of glomerular filtration flow (according clearance MDRD) or more than 100micromol plasmatic creatinine increase. 3) no renal function improvement after efficient vascular filling (>750cc normal saline or equivalent).
* Consent.

Exclusion Criteria:

* ARF not related with ATN context.
* Life expectancy less than 3 months.
* Protocol refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients experimenting ARF in ATN context.
Sampling Method: Non-Probability Sample
Enrollment: 287 (Actual)
Dates: Start 2012-04; Primary Completion 2014-10 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
PIIINP/Urinary Creatinine ratio levels between patients experimenting CRF or not. | 12months after initial diagnosis.
  We expect to highlight different ratio PIIINP/Urinary Creatinine levels and evolution between patients experimenting CRF or not (defined less than 60 mL/min according MDRD formula).

SECONDARY OUTCOMES:
NGAL/Urinary Creatinine ratio levels between patients experimenting CRF or not. | 12, 18 and 24 months after initial diagnosis.
  We expect to highlight different ratio NGAL/Urinary Creatinine levels and evolution between patients experimenting CRF or not (defined less than 60 mL/min according MDRD formula).
Correlation between NGAL/Urinary Creatinine and PIIINP/Urinary Creatinine ratios among patients with ARF. | 3, 6, 12, 18 or 24 months after initial diagnosis.
  We expect to highlight linear correlation between NGAL/Urinary Creatinine and PIIINP/Urinary Creatinine ratios among patients with ARF.
Validation of high diagnostic performance of NGAL/Urinary Creatinine ratio to predict CRF occurrence. | 3, 6, 12, 18 or 24 months after initial diagnosis.
  Sensitivity of NGAL/Urinary Creatinine ratio will be assessed at each time frame.
Validation of high diagnostic performance of PIIINP/Urinary Creatinine to predict CRF occurrence. | 3, 6, 12, 18 or 24 months after initial diagnosis.
  Sensitivity of PIIINP/Urinary Creatinine ratio will be assessed at each time frame.

IPD SHARING:
Plan to Share IPD: Undecided